CLINICAL TRIAL: NCT04900779
Title: Prospective Observational Study to Evaluate Glycocalyx Alteration in Major Abdominal and Thoracic Surgery
Brief Title: Evaluation of Glycocalyx in Major Abdominal and Thoracic Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PR(AG)569/2020
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Major Elective Abdominal and Thoracic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background:

The glycocalyx is a fundamental component of the endothelial barrier and alterations at this level have been shown to exacerbate the inflammatory response in the microcirculation. Its degradation in the surgical patient, has been tested in interventions that involve regional or general ischemia, for example in cardiac surgery, major vascular surgery or transplantation. On interventions that do not involve ischemic events the literature is limited, such is the case of those patients undergoing major abdominal and thoracic surgery.

Objective:

Assess whether there is a glycocalyx degradation in major elective abdominal and thoracic surgery, measured as an increase in plasma syndecane-1 levels during the first 24 hours of postoperative care.

Methodology:

Prospective observational study in patients undergoing major elective thoracic and abdominal surgery at the University Hospital Vall d´Hebrón. Measurement of the syndecane-1 plasma levels are going to be done during the first 24 hours after the intervention. It is intended to evaluate whether its elevation is related to anesthetic perioperative factors, and if it has an impact con morbildity and mortality in the following 6 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old
* Patients that are scheduled to major abdominal and thoracic elective surgery in Universtity Hospital Vall d´ Hebrón.
* Patients ASA I, II and III.
* Patients that after the intervention have their recovering in the Surgical ICU

Exclusion Criteria:

* Patients ASA IV and V.
* Patients that are hospitilized previous to the surgery.
* Patients that undergo emergent surgery.
* Patients with Chronic or Acute Renal Failure previous to the surgery.
* Patients with past medical history of autoinmune disseases.
* Patients with an active infection previous to the surgery.
* Patients in treatment with steroids previous to the surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years old that undergo major abdominal and thoracic elective surgery in University Hospital Vall d´Hebron.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Estimated)
Dates: Start 2021-02-02 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
plasmatic syndecan -1 levels | In the first 24 hours after the procedure
  Degradation of glucocalix measured by plasmatic syndecan -1 levels

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Vall d´Hebron, Barcelona, Spain